CLINICAL TRIAL: NCT03335566
Title: A Phase 3 Multicentre, Randomised, Comparative Study of the Efficacy and Safety of the Ultrasound Contrast Agents Sonazoid™ and SonoVue® in Subjects With Focal Liver Lesions Undergoing Pre- and Post-Contrast Ultrasound Imaging
Brief Title: An Efficacy and Safety Study of Sonazoid™ and SonoVue® in Participants With Focal Liver Lesions, Undergoing Pre- and Post-Contrast Ultrasound Imaging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-045-002; GE-045-002 (Other: GE HealthCare)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2018-08-27 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Liver Lesions
MeSH Terms: interventions — Sonazoid; contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonazoid™ (Experimental): Participants will receive single intravenous (I.V) bolus injection of Sonazoid™ 0.12 microliter (µL) microbubbles (MB)/kilogram (kg) body weight.
  Interventions: Drug: Sonazoid™
- SonoVue® (Active Comparator): Participants will receive single I.V bolus injection of SonoVue® 2.4 milliliter (mL).
  Interventions: Drug: SonoVue®

INTERVENTIONS:
Drug: Sonazoid™ — Single Dose of Sonazoid™ 0.12 µL MB/kg as I.V. injection.
  Arms: Sonazoid™
Drug: SonoVue® — Single Dose of SonoVue® 2.4 mL as I.V. injection.
  Arms: SonoVue®

SUMMARY:
The purpose of this study is to compare the efficacy of Sonazoid™ and SonoVue® in participants with focal liver lesions (FLLs), by comparing pre-and post-contrast ultrasound examination findings with regard to various aspects of lesion diagnosis including diagnosis as benign versus malignant, specific lesion diagnosis, confidence in diagnosis, and quality of delineation of lesion-related blood vessels (from images obtained during vascular imaging) and detection of lesion presence and quality of delineation of the whole liver (from images obtained during whole liver imaging).

ELIGIBILITY:
Inclusion Criteria: Participants may be included in the study if they meet all of the following criteria:

* Participant has at least 1 untreated focal liver lesions (FLL) but =<8 lesions (excluding cysts) <10 centimeter (cm) in diameter confirmed in a diagnostic examination performed in the past month (or past 3 months if lesion is benign) that can be visualised by non- contrast-enhanced (CE) ultrasound
* Participant has had a dynamic CE-computed tomography (CE-CT) or CE-magnetic resonance imaging (CE-MRI) examination within the past month or is scheduled to have one in the month following inclusion in the study and the original images (or copies thereof) are/will be available. (This inclusion criterion does not apply for participants enrolled as training cases. Investigators will be asked to submit standard of truth/ reference diagnosis for training cases whenever possible, since the cases may be used for training and testing the blinded readers prior to the blinded read)
* Participant is a 20- to 80-year-old inpatient or outpatient referred for an ultrasound examination of the liver
* Participant is able and willing to comply with study procedures and will give their signed and dated informed consent
* The participant, if female, is either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), or non-lactating, or if of childbearing potential the results of a serum or urine human chorionic gonadotropin pregnancy test, performed on the day of investigational medicinal product (IMP) administration (with the result known before IMP administration), are negative

Exclusion Criteria:

* The participant has an acute clinically fatal condition (i.e., not expected to survive for at least 6 months)
* The participant has previously received Sonazoid™ or has received SonoVue® within the past 30 days
* The participant has undergone or is undergoing systemic or loco-regional chemotherapy, or radiation therapy
* The participant is participating in another clinical trial with an unregistered medicinal product, or less than 30 days have passed since completing participation in such a trial
* The participant has a history of allergies to eggs or egg products (i.e., manifested by full body rash, respiratory difficulty, oral or laryngeal swelling, hypotension or shock)
* The participant has known hypersensitivity to sulphur hexafluoride or to any of the components of SonoVue®
* The participant has undergone or plans to undergo liver biopsy or surgery within the 24 hours before or after this examination
* The participant has undergone or plans to undergo an examination with a contrast agent (i.e., iodinated x-ray contrast agent, magnetic resonance imaging (MRI) contrast agent or another ultrasound contrast agent) within the 24 hours before or after this examination
* The participant is considered to be unsuitable to participate in the study by the investigator
* The participant is known to have a right-to-left shunt, severe pulmonary hypertension (pulmonary artery pressure >90 millimeter of mercury (mmHg) or uncontrolled systemic hypertension
* The participant has a recent acute coronary syndrome or clinically unstable ischaemic cardiac disease, including: evolving or ongoing myocardial infarction, typical angina at rest within the last 7 days, significant worsening of cardiac symptoms within the last 7 days, recent coronary artery intervention or other factors suggesting clinical instability (e.g., recent deterioration of electrocardiogram [ECG], laboratory or clinical findings), acute cardiac failure, Class III/IV cardiac failure, or severe rhythm disorders
* The participant has adult respiratory distress syndrome, severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli
* The participant has known thrombosis within the liver, portal, or mesenteric veins

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2014-05-11 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2015-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Tranquart, MD, PhD, Study Chair — GE Healthcare
Locations (18):
- China (11):
  - Peking Union Medical College Hospital, East Campus: No.1 Shuaifuyuan Wangfujing, Dongcheng, Beijing Municipality
  - Chinese PLA General Hospital, No. 28 Fuxing Road, Haidan, Beijing Municipality
  - Peking Union Medical College Hospital, West Campus: No. 41 Damucang Hutong, Xicheng, Beijing Municipality
  - The First Affiliated Hospital, Sun-Yat sen University, No. 58 Zhongshan Second Road, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Zhongshan University, No. 107 Yanjiang West Road, Guangzhou, Guangdong
  - Shanghai First Hospital, North Campus: No. 100 Haining Road, Hongkou, Shanghai Municipality
  - Shanghai First Hospital, South Campus: No.650 New Songjiang Road, Songjiang, Shanghai Municipality
  - Zhongshan Hospital Fudan University, No. 180 Fenglin Road, Xuhui, Shanghai Municipality
  - Shanghai Hua Shan Hospital, No. 12 Wulumuqi Middle Road, Xuhui, Shanghai Municipality
  - Shanghai Sixth Hospital, No. 600 Yishan Road, Xuhui, Shanghai Municipality
  - Shanghai Tenth People's Hospital, No. 301 Yanchang Middle Road, Zhabei, Shanghai Municipality
- South Korea (2):
  - Seoul National University Hospital, 101, Daehak-Ro, Jongno-Gu, Seoul
  - Seoul St Mary's Hospital, 222 Banpo-daero, Seocho-gu, Seoul
- Taiwan (5):
  - National Taiwan University Hospital - Yunlin Branch, No. 579, Sec. 2 Yunlin Road, Douliu, Yunlin County
  - National Taiwan University Hospital, No. 7 Chung-Shan South Road, Taipei
  - Mackay Memorial Hospital, No. 92, Sec. 2 Zhongshan N. Road, Taipei
  - Cathay General Hospital, No. 280 Jen-Ai Road, Sec. 4, Taipei
  - Taipei Veterans General Hospital, No. 201 Shih-Pai Road, Sec. 2, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centres in China, Korea and Taiwan. A total of 424 participants were enrolled between 11 May 2014 and 9 April 2015.
Pre-assignment Details: Participants were randomised in 1:1 ratio to receive either Sonazoid™ or SonoVue®.
Groups:
- Sonazoid™: Participants received single intravenous (I.V) bolus injection of Sonazoid™ 0.12 microliter (µL) microbubbles (MB)/kilogram (kg) body weight.
- SonoVue®: Participants received single I.V bolus injection of SonoVue® 2.4 milliliter (mL).
Period: Overall Study
Arm/Group | Sonazoid™ | SonoVue®
Started | 218 | 206
Completed | 214 | 203
Not Completed | 4 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Technical Problems | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Other than specified above | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety analysis set that included all enrolled participants who received either Sonazoid™ or SonoVue.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sonazoid™ | SonoVue® | Total
Number analyzed (Participants) | 218 | 206 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.61) | 52.2 (13.77) | 53.4 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 81 | 162
  Male | 137 | 125 | 262
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 218 | 206 | 424
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Accuracy Improvement in Post-Contrast Versus Pre-Contrast Ultrasound (US) Examination for Diagnosis of the Target Lesion as Malignant or Benign Against the Reference Diagnosis (RD)/Standard of Truth
Description: Accuracy improvement was calculated by the number of participants with improved diagnoses from the pre-contrast diagnosis to the post-contrast diagnosis divided by the total number of participants, multiplied by 100. Assessments were done by 3 blinded readers. Efficacy population which included all participants who received Sonazoid™ or SonoVue®, for whom pre-contrast & post-contrast images were recorded, & for whom there was a reference standard contrast-enhanced computed tomography (CECT)/contrast-enhanced magnetic resonance imaging (CE-MRI) examination or biopsy.
Time Frame: Pre-administration up to 15 minutes post-administration
Population: Analysis was performed on efficacy population. Here, number analysed=participants with available data for specified category.
Measure: Number; unit: percentage of participants
Groups:
- Sonazoid™: Participants received single I.V bolus injection of Sonazoid™ 0.12 µL MB/kg body weight.
- SonoVue®: Participants received single I.V bolus injection of SonoVue® 2.4 mL.
Arm/Group | Sonazoid™ | SonoVue®
Number analyzed (Participants) | 169 | 169
percentage of participants
  Reader 1: number analyzed (Participants) | 160 | 157
  Reader 1 | 18.1 | 24.2
  Reader 2: number analyzed (Participants) | 163 | 158
  Reader 2 | 22.1 | 14.6
  Reader 3: number analyzed (Participants) | 165 | 162
  Reader 3 | 17.0 | 16.7

2. Secondary Outcome: Number of Lesions Detected by Post-Contrast US Relative to Number of Lesions Detected by Pre-Contrast US (Both by Blinded Readers[BR]) and Number of Lesions Detected by Post-Contrast US (by BR) Relative to Number of Lesions Detected by RD (Investigators)
Description: For the cases that can be assessed by the blinded readers both pre- and post-contrast, differences were calculated between the Sonazoid™ and SonoVue® groups in the number of lesions detected during whole-liver imaging (post-contrast minus pre-contrast). The differences were also calculated between the Sonazoid™ and SonoVue® groups in the number of lesions (post-contrast minus reference diagnosis) detected during whole-liver imaging.
Time Frame: Pre-administration up to 15 minutes post-administration
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Lesions
Arm/Group | Sonazoid™ | SonoVue®
Number analyzed (Participants) | 169 | 169
Lesions
  Post-contrast minus Pre-contrast: Reader 1: number analyzed (Participants) | 161 | 83
  Post-contrast minus Pre-contrast: Reader 1 | 0.0 [-1.0 to 1.0] | 0.0 [-1.0 to 0.0]
  Post-contrast minus Pre-contrast: Reader 2: number analyzed (Participants) | 165 | 72
  Post-contrast minus Pre-contrast: Reader 2 | 0.0 [-2.0 to 0.0] | -1.0 [-2.0 to 0.0]
  Post-contrast minus Pre-contrast: Reader 3: number analyzed (Participants) | 162 | 47
  Post-contrast minus Pre-contrast: Reader 3 | 0.0 [-1.0 to 0.0] | -1.0 [-2.0 to 0.0]
  Post-contrast minus Reference: Reader 1: number analyzed (Participants) | 160 | 83
  Post-contrast minus Reference: Reader 1 | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 1.0]
  Post-contrast minus Reference: Reader 2: number analyzed (Participants) | 162 | 72
  Post-contrast minus Reference: Reader 2 | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 0.0]
  Post-contrast minus Reference: Reader 3: number analyzed (Participants) | 159 | 47
  Post-contrast minus Reference: Reader 3 | 0.0 [0.0 to 1.0] | 0.0 [-1.0 to 1.0]

3. Secondary Outcome: Number of Participants With Diagnostic Confidence (Evaluated by Blinded Readers) in Pre-Contrast and Post-Contrast Ultrasound Examination Results
Description: Confidence in diagnoses from the pre- and post-contrast ultrasound examinations was evaluated based on 4-point scale: 0-Unknown (cannot make a judgement on level of confidence), 1- Not confident (another examination was required), 2- Probable (Would have more confidence if another diagnostic imaging test such as MRI or CT was performed), 3- Definite (Sufficient confidence to the extent that another diagnostic imaging test such as MRI or CT was unnecessary).
Time Frame: Pre-administration up to 15 minutes post-administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sonazoid™ | SonoVue®
Number analyzed (Participants) | 169 | 169
Participants
  Reader 1: Pre-contrast: Definite (3 points) | 10 | 11
  Reader 1: Pre-contrast: Probable (2 points) | 113 | 122
  Reader 1: Pre-contrast: Not confident (1 point) | 46 | 36
  Reader 1: Pre-contrast: Unknown (0 points) | 0 | 0
  Reader 1: Post Contrast: number analyzed (Participants) | 160 | 157
  Reader 1: Post Contrast: Definite (3 points) | 57 | 54
  Reader 1: Post Contrast: Probable (2 points) | 86 | 88
  Reader 1: Post Contrast: Not confident (1 point) | 17 | 15
  Reader 1: Post Contrast: Unknown (0 points) | 0 | 0
  Reader 2: Pre-contrast: Definite (3 points) | 15 | 12
  Reader 2: Pre-contrast: Probable (2 points) | 89 | 79
  Reader 2: Pre-contrast: Not confident (1 point) | 65 | 78
  Reader 2: Pre-contrast: Unknown (0 points) | 0 | 0
  Reader 2: Post-contrast: number analyzed (Participants) | 163 | 158
  Reader 2: Post-contrast: Definite (3 points) | 116 | 103
  Reader 2: Post-contrast: Probable (2 points) | 43 | 51
  Reader 2: Post-contrast: Not confident (1 point) | 4 | 4
  Reader 2: Post-contrast: Unknown (0 points) | 0 | 0
  Reader 3: Pre-contrast: Definite (3 points) | 38 | 36
  Reader 3: Pre-contrast: Probable (2 points) | 89 | 90
  Reader 3: Pre-contrast: Not confident (1 point) | 42 | 42
  Reader 3: Pre-contrast: Unknown (0 points) | 0 | 1
  Reader 3: Post-contrast: number analyzed (Participants) | 165 | 162
  Reader 3: Post-contrast: Definite (3 points) | 130 | 117
  Reader 3: Post-contrast: Probable (2 points) | 31 | 36
  Reader 3: Post-contrast: Not confident (1 point) | 4 | 9
  Reader 3: Post-contrast: Unknown (0 points) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Accuracy Improvement in Post-contrast Versus Pre-contrast Ultrasound Examination for Lesion-Specific Diagnoses of the Target Lesion Against the Reference Diagnosis/Standard of Truth
Description: The accuracy improvement was calculated by the number of participants with improved diagnoses from the pre-contrast diagnosis to the post-contrast diagnosis divided by the total number of participants, multiplied by 100. Assessment was performed by 3 blinded readers.
Time Frame: Pre-administration up to 15 minutes post-administration
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sonazoid™ | SonoVue®
Number analyzed (Participants) | 169 | 169
percentage of participants
  Reader 1: number analyzed (Participants) | 160 | 157
  Reader 1 | 11.9 | 21.7
  Reader 2: number analyzed (Participants) | 163 | 158
  Reader 2 | 16.6 | 15.2
  Reader 3: number analyzed (Participants) | 165 | 162
  Reader 3 | 15.8 | 19.1

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from administration of investigational medicinal product (IMP) up to the 72 hours post injection regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened any time during or after administration of IMP. Analysis was performed on safety population which included all enrolled participants who received either Sonazoid™ or SonoVue®.
Arm/Group | Sonazoid™ | SonoVue®
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/206
Serious Adverse Events (participants affected / at risk) | 0/218 | 0/206
Other Adverse Events (participants affected / at risk) | 0/218 | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.